CLINICAL TRIAL: NCT06760234
Title: Prediction of Pancreatic Cancer Prognosis Using a Multimodal Deep Learning Model Based on Intratumoral Immune Microenvironment
Brief Title: Multimodal Deep Learning Model Predicts Pancreatic Cancer Prognosis
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); Hangzhou Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: PCPAI
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Deep Learning Model; Pancreatic adenocarcinoma; prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training Cohort: Patients diagnosed with pancreatic cancer who underwent surgery and other treatments at the Second Affiliated Hospital, Zhejiang University School of Medicine
  Interventions: Diagnostic Test: No Interventions
- Test Cohort: Patients diagnosed with pancreatic cancer who underwent surgery and other treatments at the Fourth Affiliated Hospital, Zhejiang University School of Medicine and Hangzhou Hosptial of Traditional Chinese Medicine
  Interventions: Diagnostic Test: No Interventions

INTERVENTIONS:
Diagnostic Test: No Interventions — The high-throughput extraction of quantitative image features from medical images
Diagnostic Test: No Interventions — Immunohistochemical analysis

SUMMARY:
This study describes the development and validation of a deep learning prediction model, which extracts deep learning features from preoperative enhanced CT scans and analyzes postoperative pathological specimens of pancreatic cancer patients. The aim is to predict patient prognosis and response to chemotherapy treatment.

DETAILED DESCRIPTION:
This study retrospectively collected enhanced CT scan data, pathological paraffin blocks, and clinical data from pancreatic cancer patients who underwent surgery at multiple centers between March 2013 and May 2024. The pathological paraffin blocks were stained using immunohistochemistry for prognostic immune microenvironment markers, and patients were classified based on these results. Subsequently, deep learning features were extracted from enhanced CT scans, and a multimodal prediction model was constructed using imaging features and clinical information. The model's performance was evaluated using metrics including area under the receiver operating characteristic curve (AUC), accuracy, sensitivity, and specificity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pancreatic cancer, diagnosed through pathology;
2. Patients underwent surgery and received adjuvant chemotherapy after surgery.

Exclusion Criteria:

1. Missing or inadequate quality of CT,
2. Incomplete clinical or pathological data.
3. Multiple primary malignancies;
4. History of malignancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer patients who were undergo surgery and received adjuvant chemotherapy after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2026-01-03 (Actual)

PRIMARY OUTCOMES:
Performance of deep learning model | Baseline treatment
  The model's performance was evaluated using metrics including area under the receiver operating characteristic curve (AUC), accuracy, sensitivity, and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Yulian Wu, PhD., Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- the Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan Y, Du B, Pu K, Sun Y, Lv C, Hu S, Song T, Wu R, Chen Y, Tang J, Zhong Y, Bian W, Wu J, Zhang H, Ding Y, Xu H, Wu Y, Li X. Noninvasive evaluation and clinical value prediction of tumor-infiltrating neutrophil-to-T-cell ratio in pancreatic ductal adenocarcinoma. NPJ Digit Med. 2026 Jan 3. doi: 10.1038/s41746-025-02303-9. Online ahead of print. PMID 41484243